CLINICAL TRIAL: NCT05662267
Title: Targeted Trial Emulation of Kidney Alone Versus Islet-After-Kidney in Type 1 Diabetic Transplant Recipients : a French Nationwide Cohort Study
Brief Title: Kidney Alone Versus Islet-After-Kidney in Type 1 Diabetic Kidney Transplant Recipient.
Acronym: KA-IAK
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Lille (Other)
Collaborators: Agence de La Biomédecine (Other Government)
Responsible Party: Sponsor
Other Study IDs: HLJ_2022_03; DEC19-483 (Other: Number register data CHU Lille)
Record Dates: First submitted 2022-12-14; First posted 2022-12-22 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: type1diabetes; Renal Failure; End Stage Renal Disease
Keywords: Type 1 Diabetes; Pancreatic Islet Transplantation; Kidney Transplantation
MeSH Terms: conditions — Renal Insufficiency; Kidney Failure, Chronic; Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Islet-after-kidney group: Patients with type 1 diabetes with a kidney transplant received or not an islet transplantation after kidney transplantation. As soon as they received an islet transplantation, they belong to the "Islet-after-kidney group".
- Kidney alone group: Patients with type 1 diabetes with a kidney transplant who did not receive an islet transplantation belong to the " Kidney alone group ".
  Interventions: Other: Pancreatic islet transplantation after kidney transplantation

INTERVENTIONS:
Other: Pancreatic islet transplantation after kidney transplantation — Pancreatic islet transplantation consists in the intrahepatic transplantation of pancreatic islets, as a result of enzymatic digestion of a deceased-donor pancreas.
  Groups: Kidney alone group

SUMMARY:
Islet transplantation is associated with a benefit on glycaemic control compared to optimized insulin therapy in recent clinical trials. However, there is a lack of evidence concerning the long-term impact of islet transplantation on type 1 diabetic kidney transplant recipients' prognosis. The objective of the study is to assess the impact of islet transplantation in patients with type 1 diabetes and a kidney transplantation on the risk of graft failure. Every type 1 diabetic recipient transplanted with a kidney in France between 2000 and 2017 is included. Patients transplanted with pancreatic islets are compared to controls treated with insulin alone according to a matching method based on time-dependent propensity scores which allow to ensure patients comparability at the time of islet transplantation. Time-dependent propensity scores are built according to variables associated with both the probabilities of being transplanted with islets and the outcome of interest. These variables are assessed by a direct acyclic graph. The primary outcome consists in death-uncensored graft survival, defined by death or return to dialysis. Secondary outcomes include the risk of death, or the risk of death-censored graft survival.

ELIGIBILITY:
Inclusion Criteria:

* Patient is aged over 18
* With type 1 diabetes
* With End-Stage Renal disease
* Transplanted with a kidney
* Between 2000 and 2017

Exclusion Criteria:

* Patients with type 2 diabetes
* Patients with a previous pancreatic transplantation with a pancreatic graft functioning at the time of kidney transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: French patients with type 1 diabetes, transplanted between 2000 and 2017 with a kidney transplant
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-03-10 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Graft failure defined by death-uncensored graft survival, i.e. the return to dialysis or death | From the date of islet transplantation (or time-point equivalent in the control group) until the date of death from any cause or return to dialysis, whichever comes first, assessed up to 240 months.

SECONDARY OUTCOMES:
Patient survival | From the date of islet transplantation (or time-point equivalent in the control group) until the date of death from any cause, assessed up to 240 months
Death-censored graft survival | From the date of islet transplantation (or time-point equivalent in the control group) until the date of death from any cause, assessed up to 240 months

CONTACTS AND LOCATIONS:
Overall Officials: Medhi Maanaoui, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hop Claude Huriez Chu Lille, Lille, France